CLINICAL TRIAL: NCT03762980
Title: Effect of Bilateral Training for Upper Extremities in Chronic Stroke Patients
Brief Title: "Bilateral Training in Stroke Patients"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shifa International Hospital (Other)
Responsible Party: Principal Investigator, Humera Ambreen, Bilateral training in stroke patients, Shifa International Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 563-011-2016
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right hemiplegic patients (Experimental)
  Interventions: Other: Bilateral training (BAT)
- Left hemiplegic patients (Experimental)
  Interventions: Other: Bilateral training (BAT)

INTERVENTIONS:
Other: Bilateral training (BAT) — Each group received bilateral training) for upper extremities for 3 days per week for 01 hour/day for up to 6 weeks. Tasks included functional tasks such as stacking cones and cups, positioning the cup upright, throw a ball into basket, carrying a wooden block and buttoning and unbuttoning of shirt with counting. Each task was performed for 10 minutes and had a rest break of 1 minute.

SUMMARY:
The objective of this study was to evaluate the effects of bilateral training for upper extremity in stroke patients and to compare these effects between right and left stroke patients. A Quasi Experimental Study conducted on community stroke survivors. A total of 24 stroke patients were included and divided into Group A (Right hemiplegia) (n=12) and Group B (Left hemiplegia) (n=12). Chronic stroke patients (>3 months), aged 30-70 years with left or right sided diagnosed stroke patients were included while patients on medication that could affect the cognitive functions or with any other cognitive impairments who are not able to follow commands were excluded. Both groups received the same intervention of with bilateral arm training involving 5 functional tasks to improve the functional activities of daily living in upper extremities. Fugl-Meyer Assessment-Upper Extremity Tool (FMA-UE) and Wolf-Motor Function Test (WMFT) were used to assess as outcome measures.The measurements were obtained at baseline and after 6th week of training. Data was analyzed using SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:

* left or right-sided chronic stroke patients

Exclusion Criteria:

* Patients with cognitive impairment or unable to follow commands

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Wolf Motor Function Test | 6 weeks
  The Wolf Motor Function Test (WMFT) was used to assess upper extremity (UE) motor ability through timed and functional tasks
Fugl Meyer Assessment-upper Extremity | 6 weeks
  Used to measure upper limb sensorimotor function in stroke patients

IPD SHARING:
Plan to Share IPD: Undecided